CLINICAL TRIAL: NCT04648852
Title: Heart Failure Burden and Heart Failure Risk in the General Population in Norway: "The HUNT for Heart Failure" Risk Score
Brief Title: The HUNT for Heart Failure" Risk Score
Acronym: HUNT4HF
Status: Completed | Type: Observational
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Boehringer Ingelheim (Industry); Norwegian University of Science and Technology (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: LH-20H4HF
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
Keywords: risk factor; population; diagnosis; prognosis
MeSH Terms: conditions — Heart Failure; Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Biobank available, but not included in this project. Laboratory test made available are haematology overview, renal function serology, C-reactive protein
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants in the third wave of the HUNT study: General population participating in the third wave of the HUNT study
  Interventions: Other: Heart failure risk estimation
- Participants in the second wave of the HUNT study: General population participating in the second wave of the HUNT study
  Interventions: Other: Heart failure risk estimation

INTERVENTIONS:
Other: Heart failure risk estimation — Evaluation by heart failure risk score

SUMMARY:
In this population study aim is to evaluate risk factors for heart failure and combine these into a new heart failure risk score.

Secondly, the heart failure risk score will be internally and externally validated, and compared with established heart failure risk scores. Additionally, the prevalence of heart failure as well as the distribution of the heart failure risk score in the general population will be evaluated.

DETAILED DESCRIPTION:
Explore which clinical risk factors or patient characteristics in a general population that are associated with increased risk for heart failure events and combine these into a new population-based heart failure risk score ("The HUNT for heart failure risk score") for predicting heart failure risk

Validate the newly developed heart failure risk score internally in the HUNT2 database

Compare the predictive ability of the new heart failure risk score with established heart failure risk scores (the ABC Health HF risk score, the Framingham HF risk score) and an established Norwegian cardiovascular risk score (NORRISK 2)

Estimate the prevalence of likely ("undiagnosed") heart failure , i.e., patients at high risk of HF, in a general population by using both the established heart failure risk scores and the newly developed heart failure risk score, and compare the heart failure event rate between those at high risk of heart failure and those with established heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the third or second wave of the HUNT study

Exclusion Criteria:

* Not willing to participate
* Missing vital data

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 36511 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Time to incident heart failure event | 10 years
  Time to first heart failure hospitalization or heart failure related visit at the out-patient clinic (events defined according to the ESC 2016 heart failure guidelines)

SECONDARY OUTCOMES:
Time to death from any cause | 10 years
  Time to death from any cause
Time to first heart failure event or death from any cause | 10 years
  Time to first heart failure event (hospitalization or HF related visit at the out-patient clinic) or death from any cause
Validity of heart failure risk score | 10 years
  Evaluation of the validity of heart failure risk score

OTHER OUTCOMES:
Prevalence of heart failure | 0 days
  Prevalence of heart failure in a general population
Distribution of heart failure risk score categories | 0 days
  Distribution of the heart failure risk score categories in a general population

CONTACTS AND LOCATIONS:
Overall Officials: Håvard Dalen, MSc, PhD, Study Chair — Helse Nord-Trøndelag HF
Locations (1):
- Levanger hospital, Levanger, Norge, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Will follow the institutional regulations

REFERENCES:
- [Derived] Ofstad AP, Brunborg C, Johansen OE, Morkedal B, Fagerland MW, Laugsand LE, Gullestad LL, Dalen H. Development of a tool to predict the risk of incident heart failure in a general population: the HUNT for HF risk score. ESC Heart Fail. 2023 Oct;10(5):2807-2815. doi: 10.1002/ehf2.14390. Epub 2023 May 29. PMID 37248650